CLINICAL TRIAL: NCT05593536
Title: Effect of Biological Nurturing Education to Pregnant Women on Breastfeeding Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Elif Dogan, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022/84
Record Dates: First submitted 2022-08-25; First posted 2022-10-25 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Breastfeeding
Keywords: biological nurturing; breastfeeding; education
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (biological nurturing) (Experimental): In biological feeding, the mother takes a semi-sitting position and the baby lies face down on the mother's breast and belly, with every part of her body in contact with the mother.
  Interventions: Behavioral: Breastfeeding Education
- Group 2 (classic breastfeeding) (Experimental): In classical breastfeeding, the mother holds her baby in her arms and breastfeeds while she is in a sitting position.
  Interventions: Behavioral: Breastfeeding Education
- Group 3 (control) (No Intervention): The mother will breastfeed her baby as she wishes.

INTERVENTIONS:
Behavioral: Breastfeeding Education — Biological feeding and classical breastfeeding trainings will be given to pregnant women by a trained nurse.
  Arms: Group 1 (biological nurturing); Group 2 (classic breastfeeding)

SUMMARY:
Aim: This study was randomized to determine the effect of biological nurturing education given to nulliparous pregnant women on breastfeeding status.

Method: The population of the study consisted of pregnant women who are visiting Istanbul Training and Research Hospital Suleymaniye Obstetrics and Pediatrics Hospital between October 2022 and August 2023. F test at 90% effect power 0.25 medium effect level on the sample of the study analyzed using the Gpower (3.1.9.2) Programe. As a result of the analyze, it was planned to recruit 207 nulliparous pregnant women. According to the calculation made, there should be at least 69 people in each groups. Accordingly, 69 people in the experimental 1 group (biological nurturing), 69 people in the experimental 2 group (classical breastfeeding), 69 people should be included in the control group. Experimental 1 group and experimental 2 group will be given breastfeeding training on their first visit and after two weeks. Breastfeeding success in the postpartum period will be compared in all groups.

ELIGIBILITY:
Inclusion Criteria:

GROUP 1:

* 18-35 age range
* Nulliparous Pregnancy
* Single Pregnancy
* Gestational week 34- 36
* Those who are literate
* Those who have a smart phone and have the opportunity to benefit from teaching methods

GROUP 2:

* 18-35 age range
* Nulliparous Pregnancy
* Single Pregnancy
* Gestational week 34-36
* Those who are literate

GROUP 3:

* 18-35 age range
* Nulliparous Pregnancy
* Single Pregnancy
* Gestational week 34-36 gw
* Those who are literate

Exclusion Criteria:

GROUP1:

* Presence of chronic disease
* Nipple problems
* Admission of the baby to the neonatal intensive care unit
* The presence of anomaly related to the baby (chromosomal anomaly, cleft palate/lip, tongue tie)
* Mothers in whom breastfeeding will be prohibited/suspected in the postpartum period
* The presence of a disease in the mother that will prevent breastfeeding
* Pregnant women with vision and hearing problems

GROUP 2:

* Presence of chronic disease
* Nipple problems
* Admission of the baby to the neonatal intensive care unit
* The presence of anomaly related to the baby (chromosomal anomaly, cleft palate/lip, tongue tie)
* Mothers in whom breastfeeding will be prohibited/suspected in the postpartum period
* The presence of a disease in the mother that will prevent breastfeeding
* Pregnant women with vision and hearing problems

GROUP 3:

* Pregnant women who go to pregnancy school
* Presence of chronic disease
* Nipple problems
* Admission of the baby to the neonatal intensive care unit
* The presence of anomaly related to the baby (chromosomal anomaly, cleft palate/lip, tongue tie)
* Mothers in whom breastfeeding will be prohibited/suspected in the postpartum period
* The presence of a disease in the mother that will prevent breastfeeding
* Pregnant women with vision and hearing problems

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 207 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Higher ''Prenatal Breastfeeding Self-Efficacy Scale'' score in the biological nurturing group | Two weeks after the first training
  Prenatal Breastfeeding Self-Efficacy Scale was developed to determine the breastfeeding self-efficacy perceptions of pregnant women in the prenatal period. The lowest score is 20, the highest score is 100. The higher the score, the higher the perception of breastfeeding self-efficacy.
Higher ''Prenatal Breastfeeding Self-Efficacy Scale'' score in the biological nurturing group | The first 24 hours of the postpartum period
  Prenatal Breastfeeding Self-Efficacy Scale was developed to determine the breastfeeding self-efficacy perceptions of pregnant women in the prenatal period. The lowest score is 20, the highest score is 100. The higher the score, the higher the perception of breastfeeding self-efficacy.
Higher ''LATCH Scale'' score in the biological nurturing group | The first 24 hours of the postpartum period
  LATCH Scale is an assessment tool to evaluate the effectiveness of early breast-feeding. A numerical score of 0, 1, or 2 is assigned to the five letters of the acronym: Latching of infant onto the breast, Amount of audible swallowing, Type of nipple, Comfort of mother, Help needed by mother to hold baby to breast. Lower scores (< 5) can indicate the need for assistance for better success at breast-feeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen SS, Alexander DD, Krebs NF, Young BE, Cabana MD, Erdmann P, Hays NP, Bezold CP, Levin-Sparenberg E, Turini M, Saavedra JM. Factors Associated with Breastfeeding Initiation and Continuation: A Meta-Analysis. J Pediatr. 2018 Dec;203:190-196.e21. doi: 10.1016/j.jpeds.2018.08.008. Epub 2018 Oct 4. PMID 30293638
- [Background] Wang Y, Zhao T, Zhang Y, Li S, Cong X. Positive Effects of Kangaroo Mother Care on Long-Term Breastfeeding Rates, Growth, and Neurodevelopment in Preterm Infants. Breastfeed Med. 2021 Apr;16(4):282-291. doi: 10.1089/bfm.2020.0358. Epub 2021 Feb 2. PMID 33533688
- [Background] Omidi A, Rahmani S, Amini R, Karami M. The effect of a planned lactation education program on the mother's breastfeeding practice and weight gain in low birth weight infants: a randomized clinical trial study. BMC Pregnancy Childbirth. 2022 Jun 13;22(1):482. doi: 10.1186/s12884-022-04810-z. PMID 35698072
- [Background] von Salmuth V, Brennan E, Kerac M, McGrath M, Frison S, Lelijveld N. Maternal-focused interventions to improve infant growth and nutritional status in low-middle income countries: A systematic review of reviews. PLoS One. 2021 Aug 18;16(8):e0256188. doi: 10.1371/journal.pone.0256188. eCollection 2021. PMID 34407128
- [Background] Huda MH, Chipojola R, Lin YM, Lee GT, Shyu ML, Kuo SY. The Influence of Breastfeeding Educational Interventions on Breast Engorgement and Exclusive Breastfeeding: A Systematic Review and Meta-Analysis. J Hum Lact. 2022 Feb;38(1):156-170. doi: 10.1177/08903344211029279. Epub 2021 Jul 6. PMID 34229526
- [Background] Araban M, Karimian Z, Karimian Kakolaki Z, McQueen KA, Dennis CL. Randomized Controlled Trial of a Prenatal Breastfeeding Self-Efficacy Intervention in Primiparous Women in Iran. J Obstet Gynecol Neonatal Nurs. 2018 Mar;47(2):173-183. doi: 10.1016/j.jogn.2018.01.005. Epub 2018 Feb 3. PMID 29406289
- [Background] Huang P, Yao J, Liu X, Luo B. Individualized intervention to improve rates of exclusive breastfeeding: A randomised controlled trial. Medicine (Baltimore). 2019 Nov;98(47):e17822. doi: 10.1097/MD.0000000000017822. PMID 31764775
- [Background] Lumbiganon P, Martis R, Laopaiboon M, Festin MR, Ho JJ, Hakimi M. Antenatal breastfeeding education for increasing breastfeeding duration. Cochrane Database Syst Rev. 2016 Dec 6;12(12):CD006425. doi: 10.1002/14651858.CD006425.pub4. PMID 27922724
- [Background] Moraes GGW, Christoffel MM, Toso BRGO, Viera CS. Association between duration of exclusive breastfeeding and nursing mothers' self-efficacy for breastfeeding. Rev Esc Enferm USP. 2021 May 10;55:e03702. doi: 10.1590/S1980-220X2019038303702. eCollection 2021. English, Portuguese. PMID 33978141
- [Background] Parry KC, Tully KP, Hopper LN, Schildkamp PE, Labbok MH. Evaluation of Ready, Set, BABY: A prenatal breastfeeding education and counseling approach. Birth. 2019 Mar;46(1):113-120. doi: 10.1111/birt.12393. Epub 2018 Sep 6. PMID 30191591
- [Background] Sayres S, Visentin L. Breastfeeding: uncovering barriers and offering solutions. Curr Opin Pediatr. 2018 Aug;30(4):591-596. doi: 10.1097/MOP.0000000000000647. PMID 29782384
- [Background] Milinco M, Travan L, Cattaneo A, Knowles A, Sola MV, Causin E, Cortivo C, Degrassi M, Di Tommaso F, Verardi G, Dipietro L, Piazza M, Scolz S, Rossetto M, Ronfani L; Trieste BN (Biological Nurturing) Investigators. Effectiveness of biological nurturing on early breastfeeding problems: a randomized controlled trial. Int Breastfeed J. 2020 Apr 5;15(1):21. doi: 10.1186/s13006-020-00261-4. PMID 32248838